CLINICAL TRIAL: NCT04460495
Title: Quantifying Tumor Respiration Using Oxygen-Enhanced Molecular MRI
Brief Title: Quantifying Oxygen Utilization of Tumors Using Oxygen-Enhanced Molecular MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-000449; NCI-2020-03446 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-06-15; First posted 2020-07-07 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: oxygen-enhanced molecular MRI in healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Feasibility (ASL,pH-Weighted amine CEST, O2-Weighted SAGE-EPI) (Experimental): Participants undergo ASL perfusion, pH-weighted amine CEST, and oxygen-weighted SAGE-EPI , while breathing normal room air (21% oxygen). Patients then undergo another ASL perfusion, pH-weighted amine CEST, and oxygen-weighted SAGE-EPI while breathing medical grade air (100% oxygen). Total ASL perfusion, pH-weighted amine CEST, and oxygen-weighted SAGE-EPI imaging scan time is 60 minutes.
  Interventions: Procedure: Arterial Spin Labeling Magnetic Resonance Imaging; Procedure: pH-Weighted amine CEST; Procedure: Oxygen-weighted SAGE-EPI

INTERVENTIONS:
Procedure: Arterial Spin Labeling Magnetic Resonance Imaging — Undergo ASL scan
  Other Names: ARTERIAL SPIN LABELING FUNCTIONAL MRI; Arterial Spin Labeling MRI; ASL; ASL fMRI
Procedure: pH-Weighted amine CEST — Undergo pH Weighted amine CEST
  Other Names: Amine CEST; CEST-EPI
Procedure: Oxygen-weighted SAGE-EPI — Undergo Oxygen-weighted SAGE-EPI
  Other Names: SAGE-EPI; Hypoxia MRI

SUMMARY:
This trial looks to study the safety and feasibility of using oxygen-enhanced molecular MRI to understand how cancer cells use oxygen differently than normal cells. Cancer cells tend to utilize (or not utilize) oxygen differently than normal cells. By using the oxygen-enhanced molecular MRI, researchers will be able to create spatial "maps" depicting areas of abnormal oxygen utilization unique to cancer. This type of information may be useful for diagnosing new cancers, understanding various "subtypes" of cancer that might utilize oxygen differently, or this information may be useful for evaluating new drugs that impact cancer metabolism.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety, feasibility, and sensitivity of oxygen-enhanced molecular magnetic resonance imaging (MRI) in healthy volunteers.

II. Measure oxygen-enhanced molecular MRI characteristics in human brain tumors.

OUTLINE:

Participants undergo arterial spin labeling (ASL) MRI scan and amine chemical exchange saturation transfer spin-and-gradient echo echo-planar imaging using amine proton CEST echo spin-and-gradient echo (SAGE) EPI (CEST-SAGE-EPI) while breathing normal room air (21% oxygen). Patients then undergo another ASL MRI and CEST-SAGE-EPI while breathing medical grade air (100% oxygen). Total ASL MRI and CEST-SAGE-EPI imaging scan time is 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will include persons who at the time of scans do not present with known neurological conditions that might impact tissue imaging results
* Patient participants should have suspected or pathology-confirmed diagnosis of a brain tumor (any histological subtype including brain metastases)
* All participants must be able to obtain an MRI scan and must be able to safely breathe high concentrations of oxygen

Exclusion Criteria:

* Participants with contraindications to MRI including metal implants
* Participants who are deemed not able to or not safe to breath high concentrations of oxygen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Change in pH-weighted amine CEST MRI to measure tumor acidity (MTRasym at 3ppm) before/after oxygen enrichment | Baseline and two hours after Oxygen enrichment
  Will be measured by voxel-wise t-tests via analysis of functional NeuroImages (AFNI) software between the average R2' and MTRasym during normal room air and medical grade air.
Change in oxygen-weighted SAGE-EPI to measure oxygen extraction (R2') before and after oxygen enrichment | Baseline and two hours after Oxygen enrichment
  We will perform voxel-wise t-tests via AFNI software between the average R2' and MTRasym during normal room air and medical grade air.
Tumor blood flow as measured by cerebral blood flow (CBF) from arterial spin labeling (ASL). | Baseline and two hours after Oxygen enrichment
  Change in ASL perfusion estimates of relative cerebral blood flow (CBF) before and after oxygen enrichment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Ellingson, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States